CLINICAL TRIAL: NCT04649034
Title: Personalizing The Risk Of Stroke And Silent Brain Infarct In Cardiovascular Disease
Brief Title: Intraventricular Stasis In Cardiovascular Disease
Acronym: ISBIFLOW
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: University of Salamanca (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Javier Bermejo Thomas, Head of Cardiac Imaging. Principal Investigator., Hospital General Universitario Gregorio Marañon
Other Study IDs: FIBHGM-ISBIFLOW
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dilated Cardiomyopathy; Thrombosis Cardiac; Stroke; Hypertrophic Cardiomyopathy
Keywords: Dilated cardiomyopathy; Hypertrophic cardiomyopathy; Cardiac thrombosis; Silent brain infarct; Stroke; Fluid dynamics; Intracardiac blood flow; Echocardiography; Phase contrast magnetic resonance imaging
MeSH Terms: conditions — Cardiomyopathy, Dilated; Stroke; Cardiomyopathy, Hypertrophic | interventions — Blood Coagulation Tests; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 86 patients ischemic DCM: A cohort of 86 patients with ischemic dilated cardiomyopathy in sinus rhythm and ejection fraction (EF) of LV less than 45%
  Interventions: Diagnostic Test: Doppler echocardiogram exam; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Brain magnetic resonance; Diagnostic Test: Coagulation blood test; Diagnostic Test: Holter monitoring
- 86 patients non ischemic DCM: A cohort of 86 patients with non-ischemic dilated cardiomyopathy in sinus rhythm and ejection fraction (EF) of LV less than 45%
  Interventions: Diagnostic Test: Doppler echocardiogram exam; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Brain magnetic resonance; Diagnostic Test: Coagulation blood test; Diagnostic Test: Holter monitoring
- 86 patients hypertrophic cardiomyopathy: A cohort of 86 patients with hypertrophic cardiomyopathy in sinus rhythm and ejection fraction (EF) of LV less than 55% or with an apical aneurism diagnosed in an image test
  Interventions: Diagnostic Test: Doppler echocardiogram exam; Diagnostic Test: Cardiac magnetic resonance; Diagnostic Test: Brain magnetic resonance; Diagnostic Test: Coagulation blood test; Diagnostic Test: Holter monitoring

INTERVENTIONS:
Diagnostic Test: Doppler echocardiogram exam — A complete echocardiographic study will be performed at enrollment. The echocardiographic images will be acquired as clinically recommended. The protocol will include the acquisition of 1) 2D images in parasternal axis long and short axis; 2) 2D and Doppler tissue images in the apical planes of 4, 2 and 3 chambers; 3) Pulsed, continuous and color Doppler M (DCMM) of transmitral LV flow and LV ejection; 4) 3-Chamber apical plane with and without color Doppler; and 5) 3D LV images. DCMM images will be obtained from the apical window using 4 and 5 chamber planes. Blood flow velocity will be obtained using Color and Gray mode in the 3 chamber view during 5-10 beats in apnea.
Diagnostic Test: Cardiac magnetic resonance — A cardiac MR will be acquired within 10 days after the enrollment. The protocol includes the following sequences: cine mode of short axis from LV base to apex and 2-3-4 chambers. 3D sequence of late enhancement of inversion-recovery. Images will be acquired after 3 min and 10 min of the administration of a total of 0.2 mmol / kg of Prohance®. Intraventricular thrombosis will be monitored. Phase contrast sequences in three orthogonal planes will be acquired. Morphological parameters of LV function (LVEF), contractility ("Wall Motion Score ") and sphericity index will be measured.
Diagnostic Test: Brain magnetic resonance — A brain MR will be acquired within 10 days after the enrollment. Axial, sagittal and coronal spin echo sequence in T1, axial images in diffusion sequences (DWI), enhanced spin echo T2 and FLAIR (fluid-attenuated inversion recovery) sequences shall be obtained. A cerebral infarction will be positive when finding the presence of a focal lesion of> 3 mm in diameter that meets one of these three characteristics: (1) high signal on isotropic DWI images and low signal on the apparent coefficient map Broadcast (ADC). (2) Cavitary lesion hyperintense on T2, with no signal (or low) in the FLAIR sequence. (3) Hyperintense lesion T2 / T1 hypointense with prior distribution defect known or new in a follow-up study.
Diagnostic Test: Coagulation blood test — 5 ml of peripheral blood will be obtained for assessment of prothrombotic markers at enrollment.
Diagnostic Test: Holter monitoring — At inclusion all patients will carry a Holter device for 24 hours to ensure absence of atrial fibrillation

SUMMARY:
This study is designed to quantify the ventricular stasis in patients with different forms of cardiomyopathy and at risk of stroke (ischemic, non-ischemic dilated cardiomyopathy and hypertrophic cardiomyopathy) by post-processing of 2D color Doppler echocardiography and phase contrast-magnetic resonance images in order to establish the relationship between quantitative variables of intraventricular stasis and the prevalence of silent embolic events and/or intraventricular mural thrombosis.

DETAILED DESCRIPTION:
Cardioembolic stroke is a major source of mortality and disability worldwide and blood stasis inside the heart is the main risk factor for developing intracardiac thrombosis. We have recently developed and patented a quantitative image-based method to map blood stasis within the cardiac chambers. The method is suitable for any medical imaging modality that provides time-resolved flow maps inside the heart (magnetic resonance, echocardiography, or computational-fluid-dynamic processing from anatomical CT images). The objective of the present project is to validate this certified technology in a multicentric cross-sectional clinical trial of 258 patients with different forms of cardiomyopathy with high-risk of stroke.

We will include patients with ischemic, non-ischemic dilated cardiomyopathy and hypertrophic cardiomyopathy in sinus rhythm and an echocardiogram, cardiac and cerebral MRI will be performed. Our objective is to quantify the ventricular stasis by post-processing of 2D color Doppler echocardiography and phase contrast-magnetic resonance images in order to establish the relationship between quantifiable intraventricular stasis variables and the prevalence of silent brain infarctions (SBIs) and intracavitary thrombosis determined by magnetic resonance (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Sinus rhythm.
* Meet one of the following criteria:

  * Diagnosis of non ischemic DCM and ejection fraction (EF) of LV less than 45%
  * Diagnosis of ischemic DCM and ejection fraction (EF) of LV less than 45%
  * Diagnosis of hypertrofic myocardiophathy and ejection fraction (EF) of LV less than 55% or apical aneurism diagnosed in an image test.

Exclusion Criteria:

* Implantable defibrillation or stimulation devices not compatible with MRI.
* Hemodinamically significant heart valve disease or prosthetic heart valves.
* Claustrophobia.
* Persistent of paroxysmal atrial fibrillation (AF).
* Prior history of significant carotid disease with stenosis greater than 50%.
* Full anticoagulation therapy prior to admission or indication of anticoagulation.
* Pro-thrombotic disorders (active oncology disease, coagulation disorders…)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 258 patients with diagnosis of ischemic, non ischemic dilated cardiomyopathy or hypertrophic cardiomyopathy under follow-up in the Cardiology Department of Gregorio Marañón General University Hospital, Madrid, Hospital Universitario Clínico de Salamanca and Hospital Clinic, Barcelona, who meet all of the inclusion criteria and none of the exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of a combined binary variable consisting of ventricular thrombosis or silent brain infarct detected by magnetic resonance | Within 10 days after enrollment
  The primary outcome measure will be a combined binary variable consisting of one of the following findings: ventricular thrombosis assessed by cardiac magnetic resonance or silent brain infarct detected by brain magnetic resonance

SECONDARY OUTCOMES:
Left ventricle mural thrombosis assessed by cardiac magnetic resonance imaging | Within 10 days after enrollment
  Left ventricle mural thrombosis will be assessed by contrast cardiac MRI. Early after gadolinium contrast administration (3 min), two dimensional T1-weighted fast-field-echo sequences with an inversion-recovery prepulse will be used. A long inversion time (520 ms) will be used to identify intraventricular thrombus as a LV mass with low-signal intensity surrounded by high-signal intensity structures.
Silent brain infarcts (SBI) | Within 10 days after enrollment
  SBIs diagnosis entails the presence of a focal lesion > 3 mm that meets one of the three following criteria: 1) high signal on DWI isotropic images and low signal on the map of apparent diffusion coefficient (ADC). DWI sequence allows to detecting ischemic lesions and assessing their chronology. (2) cavitary lesion hyperintense on T2, with no signal (or low) in the FLAIR sequence usually surrounded by a ring gliotic hyperintense, hypointense on T1). (3) hyperintense lesion on T2 / T1 hypointense with prior distribution defect known or new in a follow-up study. The studies will be interpreted by a neuroradiologist blinded to clinical and echocardiographic information. For the assessment of whether the brain infarct is clinically silent, a medical history and physical examination focused on neurological symptoms will be performed including for that purpose the National Institute of Health (USA) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bermejo Thomas, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (3):
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Clínico de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bermejo J, Benito Y, Alhama M, Yotti R, Martinez-Legazpi P, Del Villar CP, Perez-David E, Gonzalez-Mansilla A, Santa-Marta C, Barrio A, Fernandez-Aviles F, Del Alamo JC. Intraventricular vortex properties in nonischemic dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2014 Mar 1;306(5):H718-29. doi: 10.1152/ajpheart.00697.2013. Epub 2014 Jan 10. PMID 24414062
- [Result] Rossini L, Martinez-Legazpi P, Vu V, Fernandez-Friera L, Perez Del Villar C, Rodriguez-Lopez S, Benito Y, Borja MG, Pastor-Escuredo D, Yotti R, Ledesma-Carbayo MJ, Kahn AM, Ibanez B, Fernandez-Aviles F, May-Newman K, Bermejo J, Del Alamo JC. A clinical method for mapping and quantifying blood stasis in the left ventricle. J Biomech. 2016 Jul 26;49(11):2152-2161. doi: 10.1016/j.jbiomech.2015.11.049. Epub 2015 Nov 30. PMID 26680013
- [Result] Vermeer SE, Longstreth WT Jr, Koudstaal PJ. Silent brain infarcts: a systematic review. Lancet Neurol. 2007 Jul;6(7):611-9. doi: 10.1016/S1474-4422(07)70170-9. PMID 17582361
- [Result] Martinez-Legazpi P, Rossini L, Perez Del Villar C, Benito Y, Devesa-Cordero C, Yotti R, Delgado-Montero A, Gonzalez-Mansilla A, Kahn AM, Fernandez-Aviles F, Del Alamo JC, Bermejo J. Stasis Mapping Using Ultrasound: A Prospective Study in Acute Myocardial Infarction. JACC Cardiovasc Imaging. 2018 Mar;11(3):514-515. doi: 10.1016/j.jcmg.2017.06.012. Epub 2017 Oct 5. No abstract available. PMID 28917683
- [Result] Delgado-Montero A, Martinez-Legazpi P, Desco MM, Rodriguez-Perez D, Diaz-Otero F, Rossini L, Perez Del Villar C, Rodriguez-Gonzalez E, Chazo C, Benito Y, Flores O, Antoranz JC, Fernandez-Aviles F, Del Alamo JC, Bermejo J. Blood Stasis Imaging Predicts Cerebral Microembolism during Acute Myocardial Infarction. J Am Soc Echocardiogr. 2020 Mar;33(3):389-398. doi: 10.1016/j.echo.2019.09.020. Epub 2019 Dec 5. PMID 31813676